CLINICAL TRIAL: NCT03741244
Title: A Randomized Controlled Clinical Trial of Temozolomide Plus Apatinib in Newly Diagnosed High-grade Glioma
Brief Title: TMZ Plus Apatinib in Newly Diagnosed High-grade Glioma：RCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Xue Xiaoying, Director of Radiotherapy, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APAglio
Record Dates: First submitted 2018-11-13; First posted 2018-11-14 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-01

CONDITIONS: Glioma
Keywords: glioma; Apatinib; VEGFR-2; temozolomide
MeSH Terms: conditions — Glioma | interventions — apatinib; Temozolomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temozolomide and apatinib (Experimental): Patients have treated with postoperative concurrent chemoradiation. Then Temozolomide (150mg/m2/d d1-5 in the first cycle, followed by 200mg/m2/d d1-5 q28d) + apatinib (500mg/d QD).
  After 6 cycles,apatinib single drug maintained until progress.
  Interventions: Drug: apatinib; Drug: Temozolomide
- Temozolomide (Active Comparator): Patients were treated with postoperative concurrent chemoradiation.Then Temozolomide alone chemotherapy 6 cycles(first cycle 150mg/m2/d d1-5, later 200mg/m2/d d1-5 q28d).
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: apatinib — Apatinib is an oral small molecule antiangiogenic targeted drug developed in China. More and more studies found that antiangiogenic drugs have outstanding performance in treating glioma. From the perspective of clinical and molecular mechanism, the combination of Temozolomide and apatinib may have synergistic effect especially to TMZ insensitivity patients(MGMT gene promoter unmethylated) and poor prognosis (IDH1 wild type) population
  Other Names: antiangiogenic targeted drug
  Arms: Temozolomide and apatinib
Drug: Temozolomide — Temozolomide，alkylating agent， is the standard first-line chemotherapy of glioma.
  Other Names: TMZ

SUMMARY:
Glioma is the most common primary malignant Brain Tumor. Although the traditional treatment (surgery, radiotherapy and chemotherapy) has been actively carried out, the curative effect of High grade glioma (HGG) is still poor.On the basis of a lot of exploration, the union medication has become a hot spot. Malignant glioma has obvious neovascularization and inhibiting angiogenesis can inhibit tumor proliferation and invasion.Studies have found that inhibiting VEGFR-2 can can reduce neovascularization and inhibit tumor growth. NCCN clinical practice guidelines recommend bevacizumab(BEV) for the treatment of recurrent malignant gliomas. AVAglio＆RTOG 0825 subgroup analysis showed that TMZ combined with antiangiogenic drugs may have advantages in the first-line treatment of patients with IDH1 wild-type high grade glioma.However, some studies have shown that bevacizumab can lead to rapid deterioration due to hypoxia or phenotypic changes. So it is urgent to find new antiangiogenic drugs. Apatinib is an oral small molecule antiangiogenic targeted drug. Apatinib plus temozolomide has been shown to be effective and tolerable in recurrent glioma. So the investigators aimed to evaluate the efficacy and safety of temozolomide combined with apatinib in the new diagnosis of high-grade glioma，and to explore the new first-line treatment of HGG, especially to TMZ insensitivity patients(MGMT gene promoter unmethylated) and poor prognosis (IDH1 wild type) population. And Find out the benefit groups of the two drugs.

DETAILED DESCRIPTION:
Glioma is the most common primary malignant Brain Tumor.High grade glioma (HGG) has the characteristics of high morbidity, high relapse and high incidence of causing disability.Despite the progress in the combined treatment of surgery, radiotherapy and chemotherapy, the 2-year survival rate and 2-year non-progression survival rate were only 27.2% and 11.2%, respectively.

TMZ is the standard first-line chemotherapy, which can prolong the overall survival time and the progression-free survival time. Although TMZ has achieved satisfactory therapeutic effect since its application, the overall response rate of TMZ alone is still low which related to the methylation level of MGMT promoter.

On the basis of a lot of exploration, the union medication has become a hot spot. Malignant glioma has obvious neovascularization and inhibiting angiogenesis can inhibit tumor proliferation and invasion.

In recent years, antiangiogenic drugs have become a new treatment for malignant glioma. In recent years, studies have found that inhibiting VEGFR-2 can improve the sensitivity of glioma to TMZ chemotherapy. NCCN clinical practice guidelines recommend bevacizumab(BEV) for the treatment of recurrent malignant gliomas. Numerous clinical trials have studied the role of bevacizumab on glioma, and proved that bevacizumab can effectively prolong PFS without significant benefit to OS. AVAglio＆RTOG 0825 subgroup analysis showed that TMZ combined with antiangiogenic drugs may have advantages in the first-line treatment of patients with IDH1 wild-type high grade glioma.

However, some studies have shown that bevacizumab can lead to rapid deterioration due to hypoxia or phenotypic changes. So it is urgent to find new antiangiogenic drugs. Apatinib is an oral small molecule antiangiogenic targeted drug developed in China. As a specific vegfr-2 receptor inhibitor, apatinib plus temozolomide has been shown to be effective and tolerable in patients with recurrent glioma, but high-level evidence is still lacking. So the investigators conducted this clinical trial aimed to explore the new first-line treatment of high-grade glioma. The combination of TMZ and apatinib may have synergistic effect especially to TMZ insensitivity patients(MGMT gene promoter unmethylated) and poor prognosis (IDH1 wild type) population, as the high-level evidence is imminent.

From the perspective of molecular mechanism, A large number of studies have shown that vascular microenvironment closely related to glioma stem cell-like cells (GSLCs) and GSLCs can stimulate the proliferation by releasing VEGF to promote angiogenesis.. There was a correlation between the expression of vegfr-2 and CD133, a molecular biomarker of cancer stem cells. Therefore, CD133 may be an indirect target for the treatment of apatinib, and the therapeutic effect of apatinib may be related to the expression of CD133, not only vegfr-2. Monitoring the expression of CD133 can reflect the content of glioma stem cells on the one hand and indirectly reflect the therapeutic effect of vegfr-2 blocker apatinib on the other hand.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Pathological or cytological diagnosis of glioma (WHO Ⅲ or Ⅳ);
3. KPS score ≥ 60;
4. The expected survival period is ≥ 3 months;
5. Blood routine examination is basically normal: a. HB ≥ 90 G /L; b. the ANC ≥ 1.5 x 10^9/L; c. PLT≥ 80 x 10^9/L (without blood transfusion within 2 weeks, or G-CSF and other hematopoietic stimulator correction) ;
6. Normal liver and kidney function.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Second primary malignancy;
3. Severe lung infection;
4. with high blood pressure although treated with medication;
5. Patients with myocardial ischemia or myocardial infarction, arrhythmia (including QT interval > 440 ms) or grade II cardiac insufficiency;
6. Conditions that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
7. Abnormal coagulation function （INR>1.5 or PT>ULN+4s or APTT >1.5 ULN);
8. Haemorrhagic tendencies or being treated with thrombolysis or anticoagulation;
9. ≥CTCAE level 2 Pulmonary hemorrhage or ≥CTCAE level 3 other organ hemorrhage occurred within 4 weeks before the first administration of the study drug;
10. Arteriovenous thrombosis in 6 months prior to first administration, Such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism;
11. Small doses of warfarin(1mg/day) or heparin(80-100mg/day) is permitted unless INR ≤1.5;
12. Serious heart, lung and bone marrow impairment;
13. History of severe hypertension or cerebral hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival（PFS） | 1 year
  Record the time from the start of enrollment to the progression of disease or death.

SECONDARY OUTCOMES:
rate of 2-year Overall survival（OS） | 2 years
  Record the time from the start of enrollment to death for any reason.
Incidence of Treatment-Emergent Adverse Events | every month
  Record the toxicity reactions of hematology, digestive tract, skin and cardiovascular system every month,Adverse reactions were classified As "WHO classification criteria for common toxic reactions of anticancer drugs".

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ying Xue, Xue, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- the Second Hospital of Hebei Medical University, Shijiazhuang, China